CLINICAL TRIAL: NCT00419393
Title: An Open-label, Long Term Follow-up Study With Keppra XR (Levetiracetam XR) for Treatment of Partial-onset Seizures
Brief Title: Long Term Follow-up Study With Keppra XR (Levetiracetam XR) for Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01281; 2007-000899-17 (EudraCT Number)
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2011-06

CONDITIONS: Epilepsy
Keywords: Keppra XR; Levetiracetam XR; long term; partial seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Keppra XR (Levetiracetam XR) (Experimental): 1000 - 3000 mg/day Keppra XR (Levetiracetam XR), flexible dosing, throughout the duration of the study (planned: approximately 6 months-3 years)
  Interventions: Drug: Keppra XR (Levetiracetam XR)

INTERVENTIONS:
Drug: Keppra XR (Levetiracetam XR) — 500 mg tablets, 1000 - 3000 mg/day, flexible dosing for duration of the study (planned: approximately 6 months-3 years).
  Other Names: Keppra XR

SUMMARY:
To provide continued treatment of Keppra XR (Levetiracetam XR) and to assess the long term safety of Keppra XR in subjects with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were randomized into study N01280 [NCT00419094], and completed the 2 week up titration period

Exclusion Criteria:

* Subjects who did not meet the inclusion/exclusion criteria for N01280 [NCT00419094]
* Subjects who were discontinued prior to the end of titration period

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, MD, Study Director — +1 877 822 9493 (UCB)
Locations (35):
- United States (16):
  - Dothan, Alabama
  - Northport, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Loxahatchee Groves, Florida
  - Atlanta, Georgia
  - Suwanee, Georgia
  - Witchita, Kansas
  - Detroit, Michigan
  - Camden, New Jersey
  - Buffalo, New York
  - Cedarhurst, New York
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - San Antonio, Texas
- Mexico (5):
  - Aguascalientes
  - Guadalajara
  - Guadalajara Jalisco
  - Mexico City
  - Monterrey
- Poland (8):
  - Bialystok
  - Gdansk
  - Katowice
  - Lodz
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
- Russia (6):
  - Kalingrad
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Samara
  - Yaroslavl

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began December 2007 recruiting in the United States, Poland, Mexico, and the Russian Federation. The study completed March 2010.
Period: Overall Study
Arm/Group | Keppra XR (Levetiracetam XR)
Started | 190 (One subject did not receive medication)
Completed | 166
Not Completed | 24
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 7
Not completed — Other: Sponsor request | 3
Not completed — Other: Subject had temporal lobectomy | 1
Not completed — Other: Site closure | 1
Not completed — Other: Other health problems | 1
Not completed — Other: Investigator decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Keppra XR (Levetiracetam XR)
Number analyzed (Participants) | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40
  Between 18 and 65 years | 147
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.44 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 79
Region of Enrollment [Number; unit: participants]
  United States | 26
  Mexico | 49
  Poland | 59
  Russian Federation | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced at Least 1 Treatment Emergent Adverse Event During the Actual Treatment Period (6 Months-2 Years)
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Time Frame: Duration of the Treatment Period (6 months-2 years)
Population: Of the 190 subjects beginning the study, 189 received at least one dose of study medication, placing them in the Safety Set (SS) analyzed here.
Measure: Number; unit: number of subjects
Groups:
- Keppra XR: 1000 - 3000 mg/day Keppra XR (Levetiracetam XR), flexible dosing, throughout the duration of the study (planned: approximately 6 months-3 years)
Arm/Group | Keppra XR
Number analyzed (Participants) | 189
number of subjects | 126

2. Primary Outcome: Number of Subjects Who Experienced at Least 1 Serious Treatment Emergent Adverse Event During the Actual Treatment Period (6 Months-2 Years)
Description: A serious adverse event is any untoward medical occurrences in a subject administered study treatment, whether or not the event is related to treatment, with at least one of the follow outcomes: death, life-threatening, initial inpatient hospitalization or prolongation of hospitalization, significant or persistent disability/incapacity, congenital anomaly/birth defect, or an important medical event that may jeopardize the subject and require a medical/surgical intervention.
Time Frame: Duration of the Treatment Period (6 months-2 years)
Population: as for outcome 1
Measure: Number; unit: number of subjects
Arm/Group | Keppra XR
Number analyzed (Participants) | 189
number of subjects | 22

3. Primary Outcome: Number of Subjects Prematurely Discontinuing Due to a Treatment-emergent Adverse Event During the Actual Treatment Period
Description: as for outcome 1
Time Frame: Duration of the Treatment Period (6 months-2 years)
Population: as for outcome 1
Measure: Number; unit: number of subjects
Arm/Group | Keppra XR
Number analyzed (Participants) | 189
number of subjects | 5

4. Secondary Outcome: Percentage of Subjects Remaining on Keppra XR Monotherapy From Study Entry Through 6 Months
Description: Among subjects in the Efficacy (EFF) population entering the study on Keppra XR monotherapy and exposed for at least 6 months, is the percentage of subjects remaining on monotherapy treatment for at least 6 months.
Time Frame: Study entry through 6 months
Population: Of the 190 subjects beginning the study, 139 are in the Efficacy (EFF) population, entered the study on Keppra XR monotherapy, and have been exposed to treatment for at least 6 months. The Efficacy population includes subjects that are in the Safety Set (SS) with at least one reported efficacy measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Keppra XR
Number analyzed (Participants) | 139
percentage of subjects | 77.0

5. Secondary Outcome: Percentage of Subjects Remaining on Keppra XR Monotherapy From Study Entry Through 12 Months
Description: Among subjects in the Efficacy (EFF) population entering the study on Keppra XR monotherapy and exposed for at least 6 months, is the percentage of subjects remaining on monotherapy treatment for at least 12 months.
Time Frame: Study entry through 12 months
Population: Of the 190 subjects beginning the study, 49 are in the Efficacy (EFF) population, entered the study on Keppra XR monotherapy, and have been exposed to treatment for at least 12 months. The Efficacy population includes subjects that are in the Safety Set (SS) with at least one reported efficacy measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Keppra XR
Number analyzed (Participants) | 49
percentage of subjects | 65.3

ADVERSE EVENTS:
Time Frame: Up to two years
Arm/Group | Keppra XR (Levetiracetam XR)
Serious Adverse Events (participants affected / at risk) | 22/189
Other Adverse Events (participants affected / at risk) | 57/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra XR (Levetiracetam XR) (N=189)
Angina pectoris (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Drowning (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Anticonvulsant toxicity (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Lumbar puncture headache (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4)
Aphasia (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Postictal paralysis (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy with contraceptive device (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra XR (Levetiracetam XR) (N=189)
Nasopharyngitis (Infections and infestations) | 15 (19)
Influenza (Infections and infestations) | 14 (27)
Headache (Nervous system disorders) | 26 (57)
Somnolence (Nervous system disorders) | 15 (18)
Dizziness (Nervous system disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.